CLINICAL TRIAL: NCT03226145
Title: Reclassifying Constipation Using Magnetic Resonance Imaging Combined With High Resolution Manometry: A Validation Study And Double-Blind Crossover Trial
Brief Title: Reclassifying Constipation Using Imaging and Manometry
Acronym: RECLAIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: University College, London (Other); Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 16105
Record Dates: First submitted 2016-12-16; First posted 2017-07-21 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2019-07

CONDITIONS: Constipation - Functional; Irritable Bowel Syndrome Characterized by Constipation
MeSH Terms: interventions — Bisacodyl; Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Active Comparator): 80 Patients : 40 FC 40 IBS-C
  Will have MRI Motility and High Resolution Manometry
  Then will have:
  Bisacodyl 10mg once daily for 10 days, and matched placebo hyoscine butylbromide Buscopan 20mg three times daily for 10 days, and matched placebo
  Both agents will have their matched placebo dispensed alongside the active product of the other agent.
  All agents to be used in this study as tools for their known mechanisms of action, rather than to assess their effects.
  Interventions: Procedure: MRI Motility; Procedure: High Resolution Manometry; Drug: Bisacodyl; Drug: Hyoscine butylbromide
- Healthy Volunteers (Active Comparator): 40 HVs Will have MRI Motility and High Resolution Manometry No other interventions
  Interventions: Procedure: MRI Motility; Procedure: High Resolution Manometry

INTERVENTIONS:
Procedure: MRI Motility — MRI sequence to assess colonic motility
Procedure: High Resolution Manometry — HRM of colon to assess motility
Drug: Bisacodyl — Given as agent to monitor effect on symptoms and then to compare with motility data. Drug itself not being tested.
  Arms: Patients
Drug: Hyoscine butylbromide — Given as agent to monitor effect on symptoms and then to compare with motility data. Drug itself not being tested.
  Other Names: Buscopan
  Arms: Patients

SUMMARY:
Constipation is a common condition in which an individual suffers with hard stools which are infrequent and difficult to pass. It is poorly understood and treatment is often unsatisfactory. Many patients also experience pain whilst others do not but it is unclear why . It is believed that the pain arises from contractions in the colon, the lower part of the intestines. Some patients with constipation have weak colonic contraction but surprisingly some, particularly those with a lot of pain have strong contractions which are poorly coordinated. These patients all suffer from constipation but would are likely to need very different treatments. At present we cannot identify what type of abnormality of colonic contractions each individual patient suffers from and so are unable to give them the best treatment. This study will take advantage of two new techniques which have been recently developed. Magnetic Resonance Imaging (MRI) which will allow us to see the contractions of the colon in response to a dose of the laxative Moviprep which increases the flow of fluid into the proximal part of the colon and High Resolution Manometry (HRM) which measures the power and direction of the contraction in much more detail than ever before using a pressure sensing catheter placed into the bowel. Using these 2 techniques we will identify the pattern of contractions in 80 patients with constipation and 40 healthy controls. Participants will then enter into a controlled trial of either a drug which stimulates contractions or one which inhibits contraction. We anticipate that the pattern of contractions identified by the non-invasive MRI technique will predict which treatment will reduce their symptoms most as effectively as the more invasive HRM. If this is the case then our MRI test of colonic responsiveness could become widely used in routine clinical practice

DETAILED DESCRIPTION:
The study will involve both patients who suffer from constipation and also healthy volunteers.

There are two parts to the study. Participants with constipation will take part in both part 1 and part 2. Healthy volunteers will only take part in Part 1.

Part 1 of the study involves participants undergoing testing of their bowel function. It will involve 4 visits to the research centre. This is a validation study to compare MRI and HRM in their assessment of colonic motility. This will test 3 hypotheses: 1) MRI parameters of colonic physiology will correlate with HRM, 2) people with constipation who report greater abdominal pain and bloating will demonstrate greater colonic motility and frequency of retrograde contractions than those who report less bloating and abdominal pain, 3) MRI motility in the right colon will correlate with motility in the left colon.

Recruitment will be from hospital clinics as well as from the community by general advertisement. All assessments will be performed in NHS hospitals or Higher Education Institutions.

Once identified, potential participants will be sent an information sheet outlining their involvement. If they are happy to proceed they will be invited to attend the research unit (either Nottingham or London). On the first visit participants will be given all information required to give informed consent to take part. They will then be asked to complete questionnaires and a bowel diary to screen them. This will be for a 2 week period. The investigators will also access medical records in this time to help our assessment. They will return after this period and their diary/questionnaire will be assessed to ensure presence (constipation group) or absence (healthy control group) of bowel disorder. They will also be asked to have a blood test to ensure they have adequate renal function (necessary for the interventions) if they do not have one recorded in the last 3 months. They will also be asked to provide stool samples in this period.

If they meet the eligibility criteria following this they will be enrolled in the study.

Participants in the constipation group will then undergo a test for evacuation disorder called the balloon expulsion test. This is used in clinical practice to assess the function of the muscles used for defecation and it is thought to play a significant role in constipation overall. It involves inserting a thin catheter with a balloon which is filled with 50ml water. This provokes the feeling of needing to defecate and the patient will be asked to attempt to expel the balloon. They will be provided with a private toilet to do this and will be asked to time how long it takes. This measure will be recorded.

All participants (constipation group & healthy controls) will then undergo two tests. These are MRI and high resolution manometry. These will happen in a randomised order and will take place at least 1 week apart.

The MRI test day will be approximately 4 hours and will involve 3 sets of MRI images (each 30mins in length) and ingestion of a laxative drink to stimulate bowel movement which will then be analysed.

The Manometry recording day takes approximately 7 hours and involves an endoscopic procedure to place the manometry catheter in the bowel. Samples will also be taken from the bowel wall during this procedure. Once the catheter is placed the participant will remain in the research unit, be given a meal to consume and motility will be recorded for 4 hours (2hrs before meal and 2hrs after). They will undergo a single abdominal x-ray to record the position of the catheter in the bowel and it will be removed at the end of the day.

Following the completion of part 1, participants with constipation will proceed to part 2.

Part 2 looks at two currently used treatments - a prokinetic (bisacodyl) and a smooth muscle relaxant (buscopan).

There are 2 hypotheses that this will test: 1) (a) constipated patients with increased motility and/or increased contractions will respond better to a smooth muscle relaxant than to a stimulant prokinetic; (b) patients with hypomotility will respond better to a prokinetic, 2) There will be no difference between the performance of MRI and HRM as a predictor of clinical response.

The investigators will provide 2 capsules: A and B. One of the capsules will contain either Buscopan or Bisacodyl and the other an inert drug, the placebo. Whichever capsule is the placebo in the first 10 days trial will be replaced by the active drug in the second part. The order in which they are taken will be randomised so neither participant nor the research workers will know which active drug they are taking for each trial period.

This part of the study will involve 4 visits. At the first visit of these, the participant will be given the pills and instructions to take them. They will be asked to complete a daily symptom and bowel habit diary during the 10-day period and return these together with any unused pills at the second visit. After 2 weeks, they will be given the next set of capsules and again complete the daily diaries that they will return together with any unused pills at the end of the fourth visit . They will also be asked to complete one further questionnaire at the end of each treatment period. This will conclude the study.

A total of 120 participants (40 healthy, 40 FC, 40 IBS-C) will take part in the study and we estimate 4-6 weeks of time for the healthy volunteers and 12 weeks for the patient group.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 16 years
2. Capacity to give informed consent for participation
3. Ability to understand written and spoken English
4. For Constipation Group: Symptoms of constipation meeting Rome IV criteria for functional constipation or constipation-predominant irritable bowel syndrome
5. For Control Group: No symptoms of constipation. This will be defined as a score of 5 or less on the Cleveland Clinic Score

Exclusion Criteria:

* 1. Participation in any clinical trials in the past 3 months 2. Inability to understand written and spoken English 2.3. Pregnancy, assessed by a urinary pregnancy test, or current breastfeeding 3.4. History of significant adverse reaction or hypersensitivity, or known contra-indication to any of the medicinal products or equipment used in the study 4.5. History declared by the candidate of certain pre-existing gastrointestinal disorders, including:

  * inflammatory bowel disease
  * coeliac disease
  * cancer of the gastrointestinal tract 5.6. Any reported history of gastrointestinal resection (excluding appendicectomy or cholecystectomy) 6.7. Presence of an intestinal stoma 7.8. Causes of secondary constipation disorders (e.g. systemic sclerosis / Parkinson's disease) 9. Inability to cease use of medicines that cause constipation or alter colonic contractility (e.g. opioids, smooth muscle relaxants, tricyclic antidepressants) 8.10. Antibiotic use in the last 3 months 9.11. Comorbidity that would prevent safe adherence to the protocol (e.g. inability to lie flat, kidney disease contraindicating use of Moviprep or prucalopride) 10.12. Judgement by the PI that the candidate who will be unable to comply with the full study protocol (e.g. diabetes, severe COPD) 11.13. Contraindication to MRI or colonic manometry
  * Examples for MRI include claustrophobia, metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
  * Examples for manometry include diagnosis of previous complications of diverticular disease or previous endoscopic complications 12.14. Clinical evidence of significant pelvic organ prolapse syndromes 13.15. Inadequate screening diary following review iii. Control Group: A screening diary that records <6 complete spontaneous bowel motions in the fortnight.

iv. Constipation Group: A screening diary that records <2 or >6 complete spontaneous bowel motions in the fortnight

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
MRI Endpoint: Maximal MRI Motility Index (MMI) of the ascending colon (AC) | During MRI scan (over 3 hours)
  MRI Measure of Colonic Motility
HRM Endpoint: Percentage time occupied by cyclical propagating activity following meal | During manometry recording (over 6 hours)
  Manometry recording of colonic motility
Difference in average worst daily pain, scored on a range 1-5 between buscopan and bisacodyl intervention periods. | Over 10 day period

SECONDARY OUTCOMES:
Maximal MMI of the descending colon (DC) | During MRI scan (over 3 hours)
Whole Gut Transit | Weighted Average Position Score of MRI transit markers 24 hours after ingestion
Number of complete spontaneous bowel movements. | 10 day period whilst on intervention (prucalopride/buscopan)
  CSBM is defined as a bowel movement occurring more than 24 hours after the most recent dose of rescue therapy, where the participant perceives complete evacuation of their rectum.
Stool consistency | 10 day period whilst on intervention (bisacodyl/buscopan)
  Defined as days per week of type 1& 2 on the Bristol Stool Form Scale (that has an integer range from 1-7)
PAC-SYM Questionnaire Score | Throughout study. Baseline then at end of each 10 day intervention period.
Area Under the Curve for pressure 0-30 minute during HRM Number of High Amplitude Propagating Contractions (HAPCs) | During manometry recording ( 6 hours)
Number of High Amplitude Propagating Contractions (HAPCs) during HRM | During manometry recording ( 6 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, Principal Investigator — University of Nottingham
Locations (3):
- United Kingdom (3):
  - University of Nottingham, Nottingham, Notts
  - Queen Mary University of London, London
  - University College London, London

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Wilkinson-Smith V, Scott M, Menys A, Wiklendt L, Marciani L, Atkinson D, Sansone S, Zdanaviciene A, Coupland C, Knowles CH, Dinning P, Taylor SA, Gowland P, Hoad CL, Corsetti M, Spiller RC. Combined MRI, high-resolution manometry and a randomised trial of bisacodyl versus hyoscine show the significance of an enlarged colon in constipation: the RECLAIM study. Gut. 2024 Dec 10;74(1):35-44. doi: 10.1136/gutjnl-2024-332755. PMID 39438126